CLINICAL TRIAL: NCT04781634
Title: Study Evaluating Safety and Efficacy of CD19 and CD22 Targeted Prime CAR-T Cell in Patients With Relapsed/Refractory B-ALL
Brief Title: a Clinical Research of CD19 and CD22 Targeted Prime CAR-T Cell in Relapsed/Refractory B-ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC025
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: B-ALL
Keywords: CD19; CD22; CAR-T
MeSH Terms: interventions — Antigens, CD19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prime CAR- T cells (Experimental): Patients will be be treated with CD19 and CD22 prime CAR- T cells
  Interventions: Biological: CD19 and CD22 targeted prime CAR-T cells

INTERVENTIONS:
Biological: CD19 and CD22 targeted prime CAR-T cells — A single infusion of CD19 and CD22 prime CAR-T cells will be administered intravenously

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of CD19 and CD22 targeted prime CAR-T cells therapy for patients with relapsed/refractory B -ALL

DETAILED DESCRIPTION:
Although the anti-CD19 CAR-T cell therapies have gained significant results in patients with relapsed and refractory B-cell hematologic malignancies.

There are patients who resisted anti-CD19 CAR-T cells or with CD19 negative relapse. To make further improvement, the investigators launch such a clinical trial using CD19 and CD22 targeted prime CAR-T cells for patients with relapsed and refractory B-ALL to evaluate the efficacy and safety of CD19 and CD22 targeted prime CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Diagnose as Relapsed and Refractory B -ALL, and meet one of the following conditions:

   1. Failed to standard chemotherapy regimens;
   2. Relapse after complete remission, high-risk and / or refractory patients ;
   3. Relapse after hematopoietic stem cell transplantation;
3. For patients with Ph + ALL, the following conditions must be met: those who have received a standard induction chemotherapy regimen and who have not achieved complete remission after TKI treatment or have relapsed after remission (cannot tolerate TKI treatment or have contraindications to TKI treatment or the presence of TKI class) Except for drug resistant patients)
4. Evidence for cell membrane CD19 or CD22 expression
5. All genders ages: 2 to 75 years
6. The expect time of survive is above 3 months;
7. KPS>60
8. No serious mental disorders ;
9. Left ventricular ejection fraction ≥50%
10. Sufficient hepatic function defined by ALT/AST≤3 x ULN and bilirubin≤2 x ULN;
11. Sufficient renal function defined by creatinine clearance≤2 x ULN;
12. Sufficient pulmonary function defined by indoor oxygen saturation≥92%;
13. With single or venous blood collection standards, and no other cell collection contraindications;
14. Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Previous history of other malignancy;
2. Presence of uncontrolled active infection;
3. Evidence of disorder that need the treatment by glucocorticoids;
4. Active or chronic GVHD
5. The patients treatment by inhibitor of T cell
6. Pregnant or breasting-feeding women;
7. Any situation that investigators regard not suitable for attending in this study (e.g. HIV , HCVinfection or intravenous drug addiction) or may affect the data analysis.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The response rate of CD19 and CD22 prime CAR-T treatment in patients with relapse/refractory B-ALL | 6 months
  The response rate of CD19 and CD22 prime CAR-T treatment will be recorded and assessed according to the National Comprehensive Cancer Network Guideline

SECONDARY OUTCOMES:
Rate of prime CAR-T cells in bone marrow | 2 years
  Determine the rate of prime CAR-T cells in bone marrow by flow cytometry
Rate of prime CAR-T cells in peripheral blood | 2 years
  Determine the rate of prime CAR-T cells in peripheral blood by flow cytometry
Quantity of prime CAR copies in bone marrow | 2 years
  Determine the quantity of prime CAR copies in bone marrow by qPCR
Quantity of prime CAR copies in peripheral blood | 2 years
  Determine the quantity of prime CAR copies in peripheral blood by qPCR
Rate of CD19 and CD22 positive cells in Bone marrow | 1 years
  Determine the rate of CD19 and CD22 positive cells in bone marrow by flow cytometry
Levels of IL-6 in Serum | 3 months
  Serological determination of IL-6
Levels of IL-10 in Serum | 3 months
  Serological determination of IL-10
Levels of TNF-α in Serum | 3 months
  Serological determination of TNF-α
Levels of CRP in Serum | 3 months
  Serological determination of CRP
Duration of Response (DOR) of CD19 and CD22 prime CAR-T treatment in patients with refractory/relapsed B-ALL | 2 years
  DOR will be assessed from the first assessment of CR/CRi to the first assessment of recurrence or progression of the disease or death from any cause (censored)
Progress-free survival(PFS) of CD19 and CD22 targeted prime CAR-T treatment in patients with refractory/relapsed B-ALL | 2 years
  PFS will be assessed from the first prime CAR-T cell infusion to death from any cause or the first assessment of progression (censored)
Overall survival(OS) of CD19 and CD22 prime CAR-T treatment in patients with refractory/relapsed B-ALL | 2 years
  OS will be assessed from the first primeCAR-T cell infusion to death from any cause (censored)

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China; Cheng Qian, PhD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- 920th Hospital of Joint Logistics Support Force, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided